CLINICAL TRIAL: NCT01466699
Title: The Relationship of Blood Pressure Variability, Arterial Stiffness and Carotid Atherosclerosis in Beijing Residents
Brief Title: The Study of Blood Pressure Variability to Impact Arterial Stiffness and Carotid Atherosclerosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Yan Li (Other)
Responsible Party: Sponsor-Investigator, Yan Li, Principal Investigator, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: WS1916673
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate whether and what extent blood pressure variability is associated with arterial stiffness and carotid atherosclerosis, furthermore to compare the difference in the relationship of the types of blood pressure variability with arterial stiffness and carotid atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Can step by himself/herself

Exclusion Criteria:

* Cardiovascular and cerebrovascular diseases
* Secondary hypertension
* Chronic cardiac, renal, gastro-intestinal, pulmonary or any other systemic disease process requiring chronic intake of prescription medications

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in this study are community residents from Being in China
Sampling Method: Probability Sample
Enrollment: 1235 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)